CLINICAL TRIAL: NCT05382845
Title: Are There Associations Between the Outcomes of Pain Provocation Tests Early in Pregnancy and the Development of Pregnancy Related Pelvic Girdle Pain?
Brief Title: Screening for Pregnancy Related Pelvic Girdle Pain
Acronym: PPGP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge County Council Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Titti (Stina) Lilje, Principal Investigator, Blekinge County Council Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BlekingCCH
Record Dates: First submitted 2022-03-23; First posted 2022-05-19 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Pain Measurement

STUDY DESIGN:
Intervention Model Description: Prediction modelling, where risk factors such as earlier trauma to the pelvis, earlier low back pain, earlier pregnancy related pelvic girdle pain, physically demanding job, contraception and the outcomes of the pain provocation tests will predict to what degree a woman is at risk of developing symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women without symptoms of pregnancy related pelvic girdle pain (Other): There is only one arm in this study. The intervention consists of tests to rule out ongoing pelvic pain, manual pain provocation tests, and questionnaire.
  Interventions: Diagnostic Test: Manual pain provocation tests

INTERVENTIONS:
Diagnostic Test: Manual pain provocation tests — Validated and empirical pain provocation tests of the pelvic joints will be performed, both to exclude ongoing symptoms, and to diagnose one or several dysfunctions. The participants will be asked questions regarding previous symptoms, traumas, type of profession etc.
  Other Names: Questionnaire

SUMMARY:
To perform clinical manual pain provocation tests of the pelvic joints in pain free pregnant women early in pregnancy, follow them until delivery, and compare those who develop PPGP with those who don't.

DETAILED DESCRIPTION:
One arm study:

Pregnant women are informed about the study at their first visit in Maternity care. Those that are interested in participating sign an informed consent, and book an appointment with a manual therapist. During the appointment five pain provocation tests are performed to the pelvic joints, and about 13 questions regarding previous low back pain, trauma to the pelvic, or pelvic pain during previous pregnancies, number of previous pregnancies, number of years with contraception, any presence of lactosis intolerance, profession, degree of physical exercises, gestational week, age, and BMI are asked by the therapist. Each participant is given a telephone call after delivery, to ask whether any pelvic pain ocurred or not, and whether sick-leave was necessary.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women before gestational week 20 without any ongoing symptoms of pain from their pelvic joints.

Exclusion Criteria:

* Fibromyalgia
* sick-leave
* working at home
* treatment of the pelvic joints during the pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — It is still not possible for other than women to become pregnant.
Enrollment: 360 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between pain provocation tests, different risk factors and full time sick-leave. | Approximately six months for each participant
  Screening of symptom free pregnant women at their first visit in Maternity care using pain provocation tests of the pelvic joints, together with known risk factors for Pregnancy related Pelvic Girdle Pain (PPGP), and a plausible association with the primary outcome full time sick-leave due to PPGP.

CONTACTS AND LOCATIONS:
Overall Officials: Stina Lilje, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- The Region Hospital of Blekinge County, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All data that other researchers may want to look at.
Supporting Information: SAP, ICF, CSR
Time Frame: 6 months after publication
Access Criteria: Upon reasonable request